CLINICAL TRIAL: NCT05888662
Title: Endo-epicardial vs Endocardial-only Catheter Ablation of Ventricular Tachycardia in Patients Withischemic Cardiomyopathy: a Randomized Controlled Study
Brief Title: Endo-epicardial vs Endocardial-only Catheter Ablation of Ventricular Tachycardia in Patients With Ischemic Cardiomyopathy (EPIC-VT)
Acronym: EPIC-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC20_9765_EPIC-VT
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Cardiomyopathy; Catheter Ablation of Ventricular Tachycardia
Keywords: ischemic cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endo-epicardial ablation (Experimental)
  Interventions: Procedure: Endo-epicardial ablation
- endocardial ablation only (Active Comparator)
  Interventions: Procedure: endocardial ablation only

INTERVENTIONS:
Procedure: Endo-epicardial ablation — Endo-epicardial ablation of ventricular tachycardia
  Arms: Endo-epicardial ablation
Procedure: endocardial ablation only — endocardial-only catheter ablation of ventricular tachycardia
  Arms: endocardial ablation only

SUMMARY:
Radiofrequency ablation of ventricular tachycardias (VTs) is the gold standard treatment of refractory VTs in patients with ischaemic heart disease. In this setting, ablation is usually performed endocardially. However, even after a procedural success there is a high risk of recurrence, particularly due to the inability to create transmural lesions. Indeed, only the endocardium of the LV has been ablated, while a significant part of the arrhythmia substrate may be located on the other side of the myocardial thickness, on the epicardial side of the LV.

First described in 1996, epicardial ablation, performed via a percutaneous subxyphoid approach, has since undergone considerable development. Electrophysiologists often use a double endo- and epicardial approach as first line therapy for the ablation of VTs complicating myocarditis or arrhythmogenic dysplasia of the right ventricle, where the substrate is most often epicardial.

For VT in ischaemic heart disease, electrophysiologists perform endocardial ablation, and often perform epicardial ablation only after several endocardial failures. Several observational studies suggest that a combined endo- and epicardial approach as first line therapy is associated with a reduced risk of VT recurrence. Since recurrent VT in patients with ischaemic heart disease as a prognostic impact in terms of morbidity and mortality, it appears essential to optimise rhythm management by ablation, by offering a combined approach from the as first approach to reduce the risk of recurrences.

The aim of our prospective, multicentre, controlled, randomized study is therefore to compare the rate of VT recurrence after ablation performed as first line therapy either by endocardial approach alone or by combined endo-epicardial approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. 1st radiofrequency ablation of VT complicating ischaemic heart disease
3. Patients with an ICD and remote monitoring
4. Having, for women of childbearing age, effective contraception until discharge from hospital
5. Have given their free and informed consent in writing
6. are affiliated to or have health insurance

Exclusion Criteria:

1. History of cardiac surgery compromising the epicardial approach (coronary artery bypass grafting, valve replacements, or other surgeries that may have caused pericardial adhesions)
2. Presence of a left intraventricular thrombus found during pre-procedure imaging
3. Anticoagulant therapy that cannot be temporarily discontinued
4. Double antiplatelet therapy that cannot be temporarily replaced by single antiplatelet therapy
5. History of pericarditis
6. Previous thoracic radiotherapy
7. Contraindication to general anaesthesia
8. Pregnant or breastfeeding woman
9. History of heparin-induced thrombocytopenia type 2 (as injection is required during the procedure)
10. Person under legal protection (safeguard of justice, curatorship, guardianship), deprived of liberty, or unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2029-10-23 (Estimated); Study Completion 2029-10-23 (Estimated)

PRIMARY OUTCOMES:
Survival free from ventricular arrhythmia recurrence | up to 5 years
  Survival free from ventricular arrhythmia recurrence, defined as the time interval between the date of ablation and the date of first ventricular arrhythmia recurrence.
  Recurrence of ventricular arrhythmia is defined as the occurrence of appropriate ICD therapy or the occurrence ventricular arrhythmia requiring hospitalisation. The occurrence of the event and the date of the event will be obtained from the ICD interrogation.
  Patients without recurrence will be censored at the date of last ICD interrogation

SECONDARY OUTCOMES:
Number of ventricular arrhythmias treated | up to 5 years
  Number of ventricular arrhythmias treated by the defibrillator with shocks or bursts of antitachycardia pacing during follow-up or the occurrence of sustained VT/VF > 30 seconds.
Percentage of patients with recurrent ventricular arrhythmia | up to 5 years
  Percentage of patients with recurrent ventricular arrhythmia
Percentage of patients with a electrical storm | up to 5 years
  Electrical storm is defined as the occurrence of at least 3 appropriate therapies (antitachycardia pacing or shocks) delivered by the defibrillator within 24 hours.
Number of serious complications | up to 5 years
  Number of serious complications related to the procedure
Number of patients hospitalized for cardiovascular reasons | up to 2 years
  Number of patients hospitalized for cardiovascular reasons (i.e. heart failure, rhythm disorders) at 2 years
Number of patients requiring a redo ablation for ventricular arrhythmia | Up to 5 years
  Number of patients requiring a redo ablation for ventricular arrhythmia
mortality rate | Up to 2 years
  2-year mortality rate
Number of patients in each group who are non-inducible at the end of the procedure | 1 day
  Number of patients in each group who are non-inducible at the end of the procedure (programmed ventricular stimulation negative)
Length of hospital stay (from surgery to return home) | Up to 2 years
  Length of hospital stay (from surgery to return home) (Day)

OTHER OUTCOMES:
Procedure duration | 1 day
  Procedure time (from puncture to catheter removal, in minutes) and duration of radiofrequency delivery (in minutes)
Percentage of patients with inappropriate therapies deliverd by the ICD | Up to 2 years
  Percentage of patients with inappropriate therapies deliverd by the ICD at 2 years
Survival free from ventricular arrhythmia recurrence according to the treatment modality | Up to 5 years
  Describe the risk of recurrence of ventricular arrhythmias according to the treatment modality (combined endoepicardial approach vs epicardial approach alone) and according to the location of the substrate (anterior vs non-anterior, septal vs non-septal, apical vs non-apical, lateral vs non-lateral, and inferior vs non-inferior).

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël MARTINS, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (12):
- France (12):
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU de Nantes, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Universitaire La Pitié-Salpêtrière - Paris, Paris
  - CHU de Rennes, Rennes
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Etienne
  - Centre Hospitalier Universitaire Toulouse - Hôtel Dieu Saint-Jacques, Toulouse
  - Centre Hospitalier Régional Universitaire Tours - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No